CLINICAL TRIAL: NCT03870438
Title: Prevention of Mother-to-child Transmission of HIV-1: Programme Evaluation and Innovative Responsive Intervention Integrated in the Expanded Programme of Immunization. PROMISE-EPI Study
Brief Title: Prevention of Mother-to-child Transmission of HIV-1 Using a Responsive Intervention
Acronym: PROMISE-EPI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: University Teaching Hospital, Lusaka, Zambia (Other); Centre Muraz (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 12397 PROMISE-EPI
Record Dates: First submitted 2019-03-04; First posted 2019-03-12 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: HIV-1
Keywords: HIV-1; PMTCT; Point of Care; PrEP; Zambia; Burkina Faso; Expanded Program of Immunization (EPI)
MeSH Terms: interventions — Lamivudine

STUDY DESIGN:
Intervention Model Description: Phase III, Randomized Control Trial, parallel, open-label, multi-country and multi-centre trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Children infected with HIV-1 will be referred to the National Programme for confirmed HIV diagnosis and immediate ART.
  For children that are not HIV-1 infected, the results on the mother's viral load will guide the next steps:
  Mothers with a detectable plasma viral load (≥ 1000 copies/mL): their children will be initiated on lamivudine oral solution.
  Mothers with an undetectable viral loads (<1000 copies/mL): their children will not be initiated on lamivudine oral solution at 6-8 weeks of age. However, additional monitoring on the viral load of the mother and the diagnosis of the child will take place at 6 months: If the maternal plasmatic viral load is ≥ 1000 copies/mL, the child will be initiated on lamivudine oral solution.
  Interventions: Drug: Lamivudine Oral Solution
- Control (No Intervention): Routine Option B+ national guidelines including HIV-1 plasmatic viral load testing will be adhered to. Visits will take place at 6-8 weeks, 6 and 12 months post-partum to collect samples from the mother for the analysis of viral load results at 12 months. In addition, at 6-8 weeks, 6 and 12 months post-partum, POC tests will be done for the diagnosis of HIV-1 in their infants (by HIV-1 DNA PCR) and results will be shared within 2 hours. Children infected with HIV-1 will be referred to the National Programme for confirmed diagnosis and immediate ART.

INTERVENTIONS:
Drug: Lamivudine Oral Solution — In the intervention arm, HIV-1 negative children with HIV-1 positive mothers who have an HIV-1 viral load ≥ 1000 copies/ml will receive lamivudine syrup orally (7.5 mg twice daily if 2 to 4 kg; 25 mg twice a day if weight <8 kg; and 50 mg twice a day if weight >8 kg). The intervention will last a maximum of 10 months (until the baby is 12 months old or until the confirmed end of breastfeeding). Breastfeeding will be considered to be ceased if the mother confirms she is no longer breastfeeding for 2 consecutive monthly visits
  Arms: Intervention

SUMMARY:
The second visit of the Expanded Programme of Immunization when the child is 2 months old (EPI-2) represents a unique opportunity to link the EPI and PMTCT programmes and to introduce preventive and therapeutic rescue interventions in order to: 1) Assess the efficacy of the PMTCT cascade up to 2 months postpartum; 2) Allow at least 80% of HIV-1-infected infants identified at the second EPI visit who were not involved in HIV care to initiate ARVs at the earliest, but no later than 2 months after confirmation of HIV diagnosis; 3) Reduce HIV-1 transmission to less than 3% between 2 and 12 months among exposed children who completed the second EPI visit

DETAILED DESCRIPTION:
In the vast majority of sub-Saharan African countries, all mothers attend an immunization (EPI) visit when their child is 6 to 8 weeks old (the first EPI visit for BCG and OPV0 vaccination, takes place at childbirth).

This study primarily aims at utilizing existing strategies to prevent postnatal HIV-1 transmission through optimizing the use of lamivudine as pre-exposure prophylaxis (PrEP) for at risk children. For this purpose, the study will use recently marketed diagnostic point of care (POC) tests at the first level of care for maternal HIV-1 viral load and early infant diagnosis (EID). This POC early infant diagnosis will also allow optimizing treatment of HIV-infected infants by offering to all the benefits of an early ART initiation.

The hypothesis is that the second visit for routine vaccination (Expanded Program of Immunization visit 2: EPI-2) represents a unique opportunity to link EPI and PMTCT programs and introduce rescue preventive and therapeutic interventions. The EPI visit will allow an opportunity to:

1. Assess the efficacy of the PMTCT cascade.
2. Identify HIV-1-infected children early and refer them for early initiation of treatment
3. Provide their children with an antiretroviral drug that can protect them from HIV-1, irrespective of their mother's adherence to ART as part of the Phase III Randomized Controlled Trial.

The Phase III RCT will be testing a rescue preventive intervention among HIV-1-uninfected children exposed to HIV-1 by their HIV-1-infected breastfeeding mothers against a control routine Option B+ implementation.

Following a brief questionnaire and counselling on ART adherence and breastfeeding, participant mothers aged 15 years or older who meet eligibility criteria will be randomized to the control or intervention arms at a 1:1 ratio.

The phase III Randomised Controlled Trial (RCT) testing a rescue preventive intervention among HIV-1-uninfected children exposed to HIV-1 by their HIV-1-infected breastfeeding mothers against a control routine Option B+ implementation.

In the control arm, routine Option B+ national guidelines including HIV-1 plasmatic viral load testing will be adhered to as part of the clinics' usual practice. Visits will take place at 6-8 weeks, 6 and 12 months post-partum to collect samples from the mother for the analysis of viral load results at 12 months. In addition, at 6-8 weeks, 6 and 12 months post-partum, POC tests will be done for the diagnosis of HIV-1 in their infants (by HIV-1 DNA PCR) and results will be shared within 2 hours. Children infected with HIV-1 will be referred to the National Programme for confirmed diagnosis and immediate ART.

The intervention arm aims at reducing the risk of HIV transmission for infants exposed to large amounts of HIV-1 through breastfeeding, which correlates with the maternal plasma viral load. At 6-8 weeks post-partum, a venous blood sample will be taken from the mothers to assess their viral load using a GenXpert® HIV RNA POC test. Concomitantly, a capillary blood sample will be taken from the child for the detection of HIV-1 (by HIV-1 DNA PCR). Children infected with HIV-1 will be referred to the National Programme for confirmed HIV diagnosis and immediate ART.

For children that are not HIV-1 infected in the intervention arm, the results on the mother's viral load will guide the next steps:

- Mothers with a detectable plasma viral load (≥ 1000 copies/mL) will receive reinforced counselling on ART adherence.

In addition, their child will be initiated on PrEP, lamivudine syrup (7.5 mg twice daily if 2 to 4 kg; 25 mg twice a day if weight <8 kg; and 50 mg twice a day if weight >8 kg). Mothers will come with their child to the study site every month (at M3, M4, M5, M7, M8, M9, M10 and M11) to collect drug supplies, safety follow-up, child's PrEP adherence adherence and counselling, mother's ART adherence and reporting. In Zambia, high risk HIV negative infants on a 12-week prophylactic regimen and are still taking ART at this visit, their first day of the study prophylaxis administration will take place at Month 3.

- Mothers with an undetectable viral loads (<1000 copies/mL) will continue receiving ART adherence counselling. However, the children of these mothers will not be initiated on PrEP on the study at 6-8 weeks of age. However, because ART compliance declines rapidly over time within the first year of initiation, additional monitoring on the viral load of the mother and the diagnosis of the child will take place at 6 months: If the maternal plasmatic viral load is ≥ 1000 copies/mL, the child will be initiated on PrEP, lamivudine syrup (7.5 mg twice daily if 2 to 4 kg; 25 mg twice a day if weight <8 kg; and 50 mg twice a day if weight >8 kg), until the baby is 12 months old or until the confirmed end of breastfeeding. Breastfeeding will be considered to be ceased if the mother confirms she is no longer breastfeeding for 2 consecutive monthly visits.

Children infected with HIV-1 will be referred to the National Programme for confirmed diagnosis and immediate ART.

ELIGIBILITY:
For HIV+ women who give consent, the measurement of their HIV-1 viral load and the detection of HIV-1 DNA in their children will be assessed.

Inclusion Criteria:

A mother/infant pair will be included in the Phase III trial if the infant:

* Is a singleton
* Is breastfed at 2 months and the mother intends to continue breastfeeding for at least 4 months (until her child is 6 months old)
* Has a negative HIV-1 PCR POC test at 2 months of age
* Has a mother who:
* Is the accompanying person to visit 2 of the EPI
* Is 15 years of age or older (in Zambia) and 20 years of age or older (in Burkina Faso) or
* If between 15 and 19 years of age (inclusive) in Burkina Faso, and is accompanied by a referent adult of her choice representing her interests and the interests of the child (parent, family member or guardian, member of an association, etc.)
* Has been confirmed to be infected with HIV-1 (with or without HIV-2)
* Has signed the consent form to participate For the mother in Zambia, the consent must be signed by herself and a witness; For the mother in Burkina Faso, the consent must be signed by herself and a witness (if illiterate) and/or a referent adult (if under 20 years of age in Burkina Faso).

For the child in Zambia, the consent must be signed by the mother. For the child in Burkina Faso, the consent must be signed by the mother and/or a referent adult (if under 20 years of age in Burkina Faso. In Burkina Faso, both parents need to sign the consent unless the mother exercises sole parental authority or if obtaining the father's consent is likely to endanger the mother and her child. In Zambia, the mother exercises sole parental authority.

Exclusion Criteria:

A mother-child couple will not be included if the child:

* Has clinical symptoms or biological abnormalities of DAIDS classification 3 or 4 for adverse events on the day of inclusion
* Has a severe congenital malformation
* Has a known allergy to the study drug or its components
* Takes emtricitabine concomitantly
* Has a mother who:
* Lives outside the study area or intending to move from the area within the next 12 months
* Is participating in another clinical trial

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — HIV-1-positive breastfeeding mothers of HIV-1-negative children (female or male)
Enrollment: 1506 (Actual)
Dates: Start 2019-12-14 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Prevention of HIV-1 transmission from HIV-1-positive mothers to their breastfeeding children | 12 months
  Postnatal HIV-1 transmission rates at 12 months in infants exposed to HIV-1 through breastfeeding

SECONDARY OUTCOMES:
Assessment of PMTCT cascade | 2 months
  Proportion of women attending the 6-8 week EPI visit who, per the records in the antenatal care clinics:
  * had attended ANC/PMTCT clinic at least once during their pregnancy
  * had been tested for HIV-1 antenatally or during childbirth
  * are HIV-1 infected Proportion of children who were HIV-1 tested with PCR at birth (Zambia only) (per the records in the antenatal care or birth clinics)
  Proportion of women with a positive HIV test who had:
  * initiated ART during pregnancy or following childbirth (per the records in the antenatal care clinics)
  * undetectable plasma viral load (<1000 HIV RNA copies/mL) as per the results obtained with the Point of Care HIV-1 PCR Viral Load in the study Proportion of babies with a positive HIV-1 PCR (as per the results obtained with the Point of Care HIV-1 PCR Qualitative in the study)
Access to ART for HIV-1 positive children | 6 months
  Proportion of HIV-infected infants identified during the second EPI visit and who were not engaged in HIV care at this time, but who will be initiated on ART within 2 months after this visit, or if infected during follow-up- within 2 months after diagnosis, (as per the results obtained with the Point of Care HIV-1 PCR Qualitative in the study)
Evaluation of the diagnostic performance of plasma HIV viral load in comparison to breastmilk viral load to identify infants at risk of transmission at 6-8 weeks, 6 months and 12 months | 6-8 weeks, 6 months, 12 months
  Proportion of plasma HIV-1 viral load levels concordant with breast milk HIV-1 viral load levels
Evaluation of the efficacy for all the participants of the intervention arm and the comparison arm sub-population following the 2020 Zambian guidelines implementation: | 12 months
  To assess the non-inferiority of a single-drug versus triple-drug prophylactic regimen to prevent HIV transmission at one year of age (HIV-transmission rate from EPI-2 visit to 12 months of age)
Evaluation of the efficacy for all the participants of the intervention arm and the comparison arm sub-population following the 2020 Zambian guidelines implementation: | 12 months
  To assess the non-inferiority of a single-drug versus triple-drug prophylactic regimen in terms of HIV-1 free survival at one year of age.
Evaluation of the safety for all the participants of the intervention arm and the comparison arm sub-population following the 2020 Zambian guidelines implementation | 12 months
  Adverse events rates at 12 months, including death and Grade 3 or 4 events on the paediatric DAIDS scale
Evaluation of the efficacy for all the participants of the intervention arm and the comparison arm sub-population before the introduction of the 2020 Zambian guidelines (including Burkina Faso control arm) | 12 months
  To assess the efficacy of a responsive intervention package to prevent HIV transmission at one year of age (HIV-transmission rate from EPI-2 visit to 12 months of age)
Evaluation of the efficacy for all the participants of the intervention arm and the comparison arm sub-population before the introduction of the 2020 Zambian guidelines (including Burkina Faso control arm) | 12 months
  To assess the efficacy of a responsive intervention package to improve HIV-1 free survival at one year of age
Evaluation of the safety for all the participants of the intervention arm and the comparison arm sub-population before the introduction of the 2020 Zambian guidelines (including Burkina Faso control arm) | 12 months
  Adverse events rates at 12 months, including death and Grade 3 or 4 events on the paediatric DAIDS scale

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Van de Perre, MD, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (6):
- Burkina Faso (2):
  - CSPS and CMA of Do and Dafra districts, Bobo-Dioulasso
  - CSPS and CMA of Baskuy and Boulmiougou districts, Ouagadougou
- Zambia (4):
  - Bauleni, Lusaka
  - Chaisa, Lusaka
  - Chilenje Level 1 hospital, Lusaka
  - Matero Main, Lusaka

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nagot N, Kankasa C, Tumwine JK, Meda N, Hofmeyr GJ, Vallo R, Mwiya M, Kwagala M, Traore H, Sunday A, Singata M, Siuluta C, Some E, Rutagwera D, Neboua D, Ndeezi G, Jackson D, Marechal V, Neveu D, Engebretsen IMS, Lombard C, Blanche S, Sommerfelt H, Rekacewicz C, Tylleskar T, Van de Perre P; ANRS 12174 Trial Group. Extended pre-exposure prophylaxis with lopinavir-ritonavir versus lamivudine to prevent HIV-1 transmission through breastfeeding up to 50 weeks in infants in Africa (ANRS 12174): a randomised controlled trial. Lancet. 2016 Feb 6;387(10018):566-573. doi: 10.1016/S0140-6736(15)00984-8. Epub 2015 Nov 19. PMID 26603917
- [Background] Mennecier A, Kankasa C, Fao P, Moles JP, Eymard-Duvernay S, Mwiya M, Kania D, Chunda-Liyoka C, Sakana L, Rutagwera D, Tassembedo S, Wilfred-Tonga MM, Mosqueira B, Tylleskar T, Nagot N, Van de Perre P; ANRS 12397 Study group. Design and challenges of a large HIV prevention clinical study on mother-to-child transmission: ANRS 12397 PROMISE-EPI study in Zambia and Burkina Faso. Contemp Clin Trials. 2021 Jun;105:106402. doi: 10.1016/j.cct.2021.106402. Epub 2021 Apr 17. PMID 33872801
- [Derived] Kankasa C, Mennecier A, Sakana BLD, Moles JP, Mwiya M, Chunda-Liyoka C, D'Ottavi M, Tassembedo S, Wilfred-Tonga MM, Fao P, Rutagwera D, Matoka B, Kania D, Taofiki OA, Tylleskar T, Van de Perre P, Nagot N; PROMISE-EPI Trial Group. Optimised prevention of postnatal HIV transmission in Zambia and Burkina Faso (PROMISE-EPI): a phase 3, open-label, randomised controlled trial. Lancet. 2024 Apr 6;403(10434):1362-1371. doi: 10.1016/S0140-6736(23)02464-9. Epub 2024 Mar 11. PMID 38484756